CLINICAL TRIAL: NCT04184336
Title: IMPACT Project Protocol: Enhanced Population-based Core Surveillance of Meningococcal Invasive Infections at Participating Centers Across Canada
Brief Title: Enhanced Population-based Core Surveillance of Meningococcal Invasive Infections at Participating Centers Across Canada
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Canadian Paediatric Society (Other)
Collaborators: Pfizer (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: MENING
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Invasive Meningococcal Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons of all ages: Persons of all ages admitted between January 1, 2016 and December 31, 2022 with a positive result of Neisseria meningitidis isolated or detected by PCR from a normal sterile site, such as blood, CSF, joint fluid, pleural, peritoneal, pericardial fluid or tissue biopsy
  Interventions: Other: surveillance

INTERVENTIONS:
Other: surveillance

SUMMARY:
Active metropolitan area surveillance for hospital admissions related to invasive infection with Neisseria meningitidis will be conducted at the 12 centers in the IMPACT network in collaboration with Public Health officials, local infection specialists and infection control practitioners during the interval from January 1, 2016 to December 31, 2022.

DETAILED DESCRIPTION:
The objectives are 3-fold, including:

1. description of affected children and adults and the nature and outcome of the infection episodes
2. incidence rate determination in defined populations, by age, serogroup and study year
3. detailed study of the organisms recovered from cases

ELIGIBILITY:
Inclusion Criteria:Neisseria meningitidis isolated or detected by PCR from a normally sterile body site or fluid, such as blood, CSF, joint fluid, pleural, peritoneal, pericardial fluid or tissue biopsy -

Exclusion Criteria:patients diagnosed based only on

1. clinical signs, gram stain, or antigen test
2. meningococci isolated only from respiratory tract, including conjunctiva, sinuses, middle ear/mastoid, throat, peritonsillar abscess, cervical lymph node, tracheal aspirate, bronchial lavage etc -

Min Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any person admitted with confirmation of an invasive meningococcal infection at all participating Centers across Canada
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Laboratory confirmed invasive meningococcal cases. | End of 2021
  Laboratory confirmed invasive meningococcal cases.

CONTACTS AND LOCATIONS:
Locations (13):
- Canada (13):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Colombia
  - Children's Hospital Research Institute of Manitoba, Winnipeg, Manitoba
  - Eastern Health Janeway Children's and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU- Sainte Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre Mere-Enfant Soleil CHU de Quebec, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - McMaster's Children Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description IMPACT public website — http://www.cps.ca/en/impact

DOCUMENTS (2):
  • Study Protocol: Study protocol (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT04184336/Prot_000.pdf
  • Study Protocol: ID_NCT04184336 (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT04184336/Prot_001.pdf